CLINICAL TRIAL: NCT01892124
Title: Healthy Hearts, Healthy Minds
Brief Title: Motivational Interviewing and Cognitive Behavioral Therapy-based Intervention for Cardiovascular Disease Prevention Amongst American Indians With Diabetic and Depressive Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Karina Walters, Professor, School of Social Work; Director, Indigenous Wellness Research Institute, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 44890-G; P60MD006909 (NIH)
Record Dates: First submitted 2013-06-28; First posted 2013-07-03 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Cardiovascular Diseases; Diabetes Mellitus, Type 2; Depression; Dysthymic Disorder
Keywords: Motivational Interviewing; Cognitive Therapy; Community-Based Participatory Research; Indians, North American
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2; Depression; Dysthymic Disorder | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Motivational Interviewing/Cognitive Behavioral-based Therapy (Experimental): Receives an immediate weekly 10 session intervention based on a culturally-adapted, motivational interviewing and Cognitive Behavioral Therapy grounded protocol.
  Interventions: Behavioral: Motivational Interviewing/Cognitive Behavioral-based Therapy
- Wait-List Control (Experimental): Receives a weekly 10 session intervention based on a culturally-adapted, motivational interviewing and Cognitive Behavioral Therapy grounded protocol after a three month, no-intervention waiting period.
  Interventions: Behavioral: Motivational Interviewing/Cognitive Behavioral-based Therapy

INTERVENTIONS:
Behavioral: Motivational Interviewing/Cognitive Behavioral-based Therapy

SUMMARY:
American Indians (AIs) living in the Northwest have very high rates of diabetes, obesity, tobacco use, depression, and other risk factors associated with cardiovascular disease. Depression and diabetes have a pernicious effect on CVD risk and susceptibility. This study seeks to build upon the success of the 1-month, 5-session motivational interviewing (MI) CVD prevention component of the həli?dxw Project (aka Healthy Hearts-originally funded under RFA-HL-06-002; U01 HL HL087322-05). həli?dxw successfully culturally adapted MI for CVD prevention for AIs, trained AIs to implement the intervention, and conducted a preliminary feasibility and efficacy trial. Initial results indicated that participants enthusiastically embraced the MI component of the program; however, observations of the counselors, survey data, and feedback from participants suggest that depressive symptomatology served as a barrier to achieving CVD preventive behaviors and desired outcomes; and, that more time and attention to underlying depressive symptomatology may enhance motivation and CVD prevention behaviors, particularly among AIs with pre-diabetes and Type 2 diabetes. Building upon solid preliminary CVD epidemiological data, preliminary acceptability and feasibility of utilizing an MI approach, and motivated by the need to address elevated depression and diabetes profiles from the həli?dxw study, the investigators will develop a 3-month, 10-session MI-based cognitive-behavioral-adherence (MI-CBT-CVD) treatment program to address underlying depressive symptomatology, activate CVD prevention behaviors, and decrease BMI and CVD risk behaviors among 50 pre-and recently diagnosed diabetic AIs at risk for CVD. The study proposes three innovative and significant aims. First, in line with community-based participatory (CBPR) principles and pre-established indigenous research protocols with the tribal community, the investigators will conduct formative research to develop the MI-CBT-CVD intervention. Second, the investigators will conduct a pilot randomized two-group, single-site waitlist-controlled clinical trial of a 10-session, 3-month MI-based cognitive-behavioral treatment for CVD prevention (MI-CBT-CVD) among 50 pre-and recently diagnosed diabetic AI adults with depressive symptomatology and who are also at risk for CVD. Assessments will be conducted at pre and post intervention and at 6-months (3 month follow-up). Third, the investigators will disseminate the findings to the tribe as well as research outlets and prepare an RO1 to conduct a full-scale RCT should the pilot intervention be efficacious, acceptable to the community, and feasible. The primary objectives will be to determine the effect of the proposed culturally-grounded behavioral intervention program on (a) reducing weight as measured by BMI (7-10% reduction in BMI); (b) decreasing depressive symptomatology; (c) increasing physical activity; (d) decreasing sedentary activities; (d) increasing healthful food habits; and (e) improving biomedical outcomes (e.g., blood lipid profiles, glucose, hemoglobin A1C, and blood pressure). The intervention will be culturally relevant and utilize existing Native resources and personnel wherever possible.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older
* Be an American Indian/Alaska Native
* Currently reside on or within 20 miles of the Tribal reservation boundary
* Have a Body Mass Index > 25
* Have a PSS (10 item) score > 15
* Be pre-diabetic for Type 2 diabetes (via self-report, health provider referral, or previous glucose reading or hemoglobin A1c reading indicating pre-diabetes within the past 12 months) or have been diagnosed as having Type 2 diabetes
* If a woman, not currently pregnant

Exclusion Criteria:

* Referred to their physician for approval of participation during the baseline assessment process and the physician does not give approval or the participant refused to follow-up on the referral
* Unstable or exhibits serious psychiatric symptoms as determined by project's tribal mental health specialist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index | Assessed at baseline, 3 month, and 6 month timepoints
  The investigators will compare changes in body mass index between the wait-list control group and the immediate intervention group, and also for each individual over time.

SECONDARY OUTCOMES:
Changes in Depressive Symptoms using the Center for Epidemiologic Studies Depression Scale (CES-D) | Assessed at baseline, 3 month, and 6 month timepoints
  The investigators will compare changes in depressive symptoms as measured by the CES-D 10-item scale between the wait-list control group and the immediate intervention group, and also for each individual over time.
Changes in Blood Lipids | Assessed at baseline, 3 month, and 6 month timepoints
  The investigators will compare changes in mg/dL of blood lipids (Total cholesterol, HDL-C, LDL-C, triglycerides) between the wait-list control group and the immediate intervention group, and also for each individual over time.
Changes in Blood Glucose | Assessed at baseline, 3 month, and 6 month timepoints
  The investigators will compare changes in mg/dL blood glucose between the wait-list control group and the immediate intervention group, and also for each individual over time.
Changes in Hemoglobin A1c | Assessed at baseline, 3 month, and 6 month timepoints
  The investigators will compare changes in percent hemoglobin A1c between the wait-list control group and the immediate intervention group, and also for each individual over time.
Changes in Blood Pressure | Assessed at baseline, 3 month, and 6 month timepoints
  The investigators will compare changes in mmHg blood pressure levels between the wait-list control group and the immediate intervention group, and also for each individual over time.

OTHER OUTCOMES:
Changes in Physical Activity | Assessed at baseline, 3 month, and 6 month timepoints
  The investigators will compare changes in physical activity levels between the wait-list control group and the immediate intervention group, and also for each individual over time.
Changes in Sedentary Activity | Assessed at baseline, 3 month, and 6 month timepoints
  The investigators will compare changes in sedentary activity levels between the wait-list control group and the immediate intervention group, and also for each individual over time.
Changes in Food Habits | Assessed at baseline, 3 month, and 6 month timepoints
  The investigators will compare changes in food habits between the wait-list control group and the immediate intervention group, and also for each individual over time.

CONTACTS AND LOCATIONS:
Overall Officials: Karina L Walters, MSW, PhD, Principal Investigator — University of Washington; Rachelle McCarty, ND, MPH, Study Director — University of Washington
Locations (1):
- University of Washington, Indigenous Wellness Research Institute, Seattle, Washington, United States

REFERENCES:
- [Background] Walters KL, LaMarr J, Levy RL, Pearson C, Maresca T, Mohammed SA, Simoni JM, Evans-Campbell T, Fredriksen-Goldsen K, Fryberg S, Jobe JB; həli?dxw Intervention Team. Project həli?dx(w)/Healthy Hearts Across Generations: development and evaluation design of a tribally based cardiovascular disease prevention intervention for American Indian families. J Prim Prev. 2012 Aug;33(4):197-207. doi: 10.1007/s10935-012-0274-z. PMID 22965622
- [Background] Mohammed SA, Walters KL, Lamarr J, Evans-Campbell T, Fryberg S. Finding middle ground: negotiating university and tribal community interests in community-based participatory research. Nurs Inq. 2012 Jun;19(2):116-27. doi: 10.1111/j.1440-1800.2011.00557.x. Epub 2011 Jul 15. PMID 22530859